CLINICAL TRIAL: NCT03182738
Title: Video Information Provider for HIV-Associated Non-AIDS (VIP-HANA) Symptoms
Acronym: VIP-HANA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Assistant Professor of Nursing, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AAAP5958; R01NR015737-01A1 (NIH)
Record Dates: First submitted 2017-05-11; First posted 2017-06-09 (Actual); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: HIV (Human Immunodeficiency Virus); AIDS (Acquired Immunodeficiency Syndrome)
Keywords: HIV/AIDS Health Management App; HIV/AIDS symptoms
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): VIP app that delivers HIV-related symptom strategies
  Interventions: Behavioral: VIP app that delivers HIV-related symptom strategies.
- Control (Sham Comparator): VIP app without HIV-related symptom strategies
  Interventions: Behavioral: VIP app without HIV-related symptom strategies.

INTERVENTIONS:
Behavioral: VIP app without HIV-related symptom strategies. — The control group will receive the VIP app without HIV-related symptom strategies
  Arms: Control
Behavioral: VIP app that delivers HIV-related symptom strategies. — The Intervention group will receive the VIP app that delivers HIV-related symptom strategies
  Arms: Intervention

SUMMARY:
The purpose of this study is to use technology to improve symptom status and ultimately improve patient centered outcomes in people living with HIV/AIDS (PLWHA). The primary purpose of the intervention (VIP-HANA) is to improve symptom status. The investigators hypothesize that VIP-HANA will improve symptom frequency and intensity.

DETAILED DESCRIPTION:
As PLWHA age, they are developing chronic illnesses and co-morbid conditions that are often seen in older HIV negative patients. HANA conditions (e.g., cardiovascular disease, liver disease, diabetes, and asthma) are becoming more common as PLWHA age.

An individual's ability to identify and self-manage symptoms of HIV illness has been shown to improve patient outcomes and quality of life. The investigators will develop and pilot test the Video Information Provider (VIP), a web application (app) that delivered HIV-related symptom self-care strategies for PLWHA for 13 common (non-HANA) HIV/AIDS symptoms. There is a need to identify the symptom experience of PLWHA with HANA conditions.

The aim is to compare the efficacy of VIP-HANA to a control arm for ameliorating symptom frequency and intensity and secondary health outcomes in 100 PLWHA with HANA conditions over 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. HIV+
2. Age 18 or over
3. Able to read and respond in English
4. Reside within the US
5. Willing to participate in an online survey.

Exclusion Criteria:

1. HIV-negative
2. under age 18
3. Unwilling to provide key data (i.e., age, information about symptoms) on the online survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University School for Nursing, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gordian-Arroyo A, Reame N, Gutierrez J, Liu J, Ganzhorn S, Igwe KC, Laing K, Schnall R. Do correlates of white matter features differ between older men and women living with human immunodeficiency virus? Menopause. 2023 Feb 1;30(2):149-155. doi: 10.1097/GME.0000000000002102. Epub 2022 Nov 20. PMID 36696639
- [Derived] Cho H, Porras T, Flynn G, Schnall R. Usability of a Consumer Health Informatics Tool Following Completion of a Clinical Trial: Focus Group Study. J Med Internet Res. 2020 Jun 15;22(6):e17708. doi: 10.2196/17708. PMID 32538796

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 50 | 50
Completed | 41 | 45
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 9 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 44 | 89
  >=65 years | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.87 (10.41) | 53.66 (11.21) | 52.77 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 27 | 44
  Male | 33 | 23 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 20 | 30
  Not Hispanic or Latino | 40 | 30 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 35 | 31 | 66
  White | 5 | 5 | 10
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 8 | 12 | 20
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Symptom Burden Score
Description: The Symptom Burden Score is an expanded version of the 20-item HIV symptom index. The score is calculated for the 28 most common symptoms in persons living with HIV. Each symptom is given a score ranging from 0 to 4 with the scores indicating the following: 0 (not experienced) , 1 (It doesn't bother me), 2 (It bothers me a little), 3 (It bothers me), or 4 (It bothers me a lot). The higher the score (closer to 4), the greater the symptom burden (worse outcome).
Time Frame: Baseline, 3 months and 6 months; period 1 = 1-6 weeks (baseline), period 2 = 6-18 weeks (3 months), period 3 = >18 weeks (6 months)
Population: The statistical analysis defined the time points into 3 periods to correlate with the baseline, 3-month, and 6-month visits. Not all participants completed the symptom burden scale and therefore did not align within the 3 designated periods.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 50 | 50
score on a scale
  Anxiety - period 1 | 1.08 (1.47) | 1.06 (1.49)
  Anxiety - period 2: number analyzed (Participants) | 42 | 46
  Anxiety - period 2 | 0.83 (1.36) | 0.71 (1.37)
  Anxiety - period 3: number analyzed (Participants) | 40 | 44
  Anxiety - period 3 | 0.80 (1.34) | 0.78 (1.38)
  Changes in appetite - period 1 | 0.85 (1.36) | 0.70 (1.19)
  Changes in appetite - period 2: number analyzed (Participants) | 42 | 46
  Changes in appetite - period 2 | 0.79 (1.34) | 0.67 (1.21)
  Changes in appetite - period 3: number analyzed (Participants) | 40 | 44
  Changes in appetite - period 3 | 0.76 (1.36) | 0.55 (1.15)
  Clumsiness or difficulty with balance - period 1 | 0.88 (1.49) | 0.82 (1.39)
  Clumsiness or difficulty with balance - period 2: number analyzed (Participants) | 42 | 46
  Clumsiness or difficulty with balance - period 2 | 0.83 (1.41) | 0.66 (1.28)
  Clumsiness or difficulty with balance - period 3: number analyzed (Participants) | 40 | 44
  Clumsiness or difficulty with balance - period 3 | 0.94 (1.49) | 0.58 (1.25)
  Difficulty concentrating - period 1 | 0.76 (1.32) | 1.14 (1.50)
  Difficulty concentrating - period 2: number analyzed (Participants) | 42 | 46
  Difficulty concentrating - period 2 | 0.68 (1.29) | 0.82 (1.37)
  Difficulty concentrating - period 3: number analyzed (Participants) | 40 | 44
  Difficulty concentrating - period 3 | 0.70 (1.31) | 0.83 (1.39)
  Constipation, gas, or bloating - period 1 | 1.28 (1.53) | 1.21 (1.47)
  Constipation, gas, or bloating - period 2: number analyzed (Participants) | 42 | 46
  Constipation, gas, or bloating - period 2 | 1.16 (1.57) | 1.11 (1.51)
  Constipation, gas, or bloating - period 3: number analyzed (Participants) | 40 | 44
  Constipation, gas, or bloating - period 3 | 1.12 (1.53) | 0.93 (1.46)
  Cough - period 1 | 0.77 (1.35) | 0.90 (1.36)
  Cough - period 2: number analyzed (Participants) | 42 | 46
  Cough - period 2 | 0.72 (1.32) | 0.76 (1.32)
  Cough - period 3: number analyzed (Participants) | 40 | 44
  Cough - period 3 | 0.76 (1.32) | 0.74 (1.29)
  Depression - period 1 | 1.36 (1.48) | 1.36 (1.62)
  Depression - period 2: number analyzed (Participants) | 42 | 46
  Depression - period 2 | 1.33 (1.58) | 1.00 (1.51)
  Depression - period 3: number analyzed (Participants) | 40 | 44
  Depression - period 3 | 1.32 (1.56) | 0.91 (1.46)
  Decreased sex drive - period 1 | 0.98 (1.49) | 1.09 (1.49)
  Decreased sex drive - period 2: number analyzed (Participants) | 42 | 46
  Decreased sex drive - period 2 | 0.85 (1.42) | 0.68 (1.32)
  Decreased sex drive - period 3: number analyzed (Participants) | 40 | 44
  Decreased sex drive - period 3 | 0.85 (1.41) | 0.58 (1.28)
  Diarrhea- period 1 | 0.81 (1.36) | 0.62 (1.19)
  Diarrhea - period 2: number analyzed (Participants) | 42 | 46
  Diarrhea - period 2 | 0.63 (1.29) | 0.52 (1.18)
  Diarrhea - period 3: number analyzed (Participants) | 40 | 44
  Diarrhea - period 3 | 0.62 (1.28) | 0.37 (0.99)
  Difficulty remembering - period 1 | 1.01 (1.45) | 1.15 (1.53)
  Difficulty remembering - period 2: number analyzed (Participants) | 42 | 46
  Difficulty remembering - period 2 | 0.92 (1.40) | 1.08 (1.51)
  Difficulty remembering - period 3: number analyzed (Participants) | 40 | 44
  Difficulty remembering - period 3 | 0.83 (1.36) | 0.97 (1.44)
  Lightheadedness or dizziness - period 1 | 0.83 (1.39) | 0.66 (1.22)
  Lightheadedness or dizziness - period 2: number analyzed (Participants) | 42 | 46
  Lightheadedness or dizziness - period 2 | 0.76 (1.35) | 0.45 (1.07)
  Lightheadedness or dizziness - period 3: number analyzed (Participants) | 40 | 44
  Lightheadedness or dizziness - period 3 | 0.82 (1.43) | 0.32 (0.91)
  Dry eyes - period 1 | 0.78 (1.30) | 0.63 (1.17)
  Dry eyes - period 2: number analyzed (Participants) | 42 | 46
  Dry eyes - period 2 | 0.63 (1.22) | 0.64 (1.18)
  Dry eyes - period 3: number analyzed (Participants) | 40 | 44
  Dry eyes - period 3 | 0.53 (1.15) | 0.57 (1.06)
  Thirst or dry mouth - period 1 | 1.35 (1.53) | 1.13 (1.41)
  Thirst or dry mouth - period 2: number analyzed (Participants) | 42 | 46
  Thirst or dry mouth - period 2 | 0.98 (1.41) | 0.96 (1.40)
  Thirst or dry mouth - period 3: number analyzed (Participants) | 40 | 44
  Thirst or dry mouth - period 3 | 0.97 (1.40) | 0.97 (1.39)
  Difficulty falling asleep - period 1 | 1.41 (1.63) | 1.52 (1.69)
  Difficulty falling asleep - period 2: number analyzed (Participants) | 42 | 46
  Difficulty falling asleep - period 2 | 1.27 (1.68) | 1.21 (1.66)
  Difficulty falling asleep - period 3: number analyzed (Participants) | 40 | 44
  Difficulty falling asleep - period 3 | 1.47 (1.74) | 1.28 (1.68)
  Fatigue - period 1 | 1.83 (1.53) | 1.73 (1.52)
  Fatigue - period 2: number analyzed (Participants) | 42 | 46
  Fatigue - period 2 | 1.41 (1.60) | 1.32 (1.51)
  Fatigue - period 3: number analyzed (Participants) | 40 | 44
  Fatigue - period 3 | 1.31 (1.53) | 1.07 (1.40)
  Fever, night sweats, or chills - period 1 | 0.72 (1.27) | 0.77 (1.40)
  Fever, night sweats, or chills - period 2: number analyzed (Participants) | 42 | 46
  Fever, night sweats, or chills - period 2 | 0.65 (1.28) | 0.63 (1.28)
  Fever, night sweats, or chills - period 3: number analyzed (Participants) | 40 | 44
  Fever, night sweats, or chills - period 3 | 0.70 (1.30) | 0.60 (1.22)
  Heartburn - period 1 | 0.96 (1.42) | 0.81 (1.44)
  Heartburn - period 2: number analyzed (Participants) | 42 | 46
  Heartburn - period 2 | 0.79 (1.34) | 0.70 (1.40)
  Heartburn - period 3: number analyzed (Participants) | 40 | 44
  Heartburn - period 3 | 0.84 (1.43) | 0.55 (1.27)
  Problems achieving an erection - period 1 | 0.72 (1.37) | 0.23 (0.83)
  Problems achieving an erection - period 2: number analyzed (Participants) | 42 | 46
  Problems achieving an erection - period 2 | 0.59 (1.25) | 0.24 (0.88)
  Problems achieving an erection - period 3: number analyzed (Participants) | 40 | 44
  Problems achieving an erection - period 3 | 0.62 (1.30) | 0.23 (0.87)
  Muscle aches or pain - period 1 | 2.17 (1.54) | 2.12 (1.59)
  Muscle aches or pain - period 2: number analyzed (Participants) | 42 | 46
  Muscle aches or pain - period 2 | 1.86 (1.59) | 1.74 (1.62)
  Muscle aches or pain - period 3: number analyzed (Participants) | 40 | 44
  Muscle aches or pain - period 3 | 1.78 (1.66) | 1.79 (1.59)
  Neuropathy - period 1 | 1.94 (1.65) | 1.67 (1.63)
  Neuropathy - period 2: number analyzed (Participants) | 42 | 46
  Neuropathy - period 2 | 1.77 (1.68) | 1.66 (1.63)
  Neuropathy - period 3: number analyzed (Participants) | 40 | 44
  Neuropathy - period 3 | 1.86 (1.64) | 1.56 (1.63)
  Pain or discomfort during sex - period 1 | 0.27 (0.87) | 0.21 (0.76)
  Pain or discomfort during sex - period 2: number analyzed (Participants) | 42 | 46
  Pain or discomfort during sex - period 2 | 0.36 (1.06) | 0.18 (0.74)
  Pain or discomfort during sex - period 3: number analyzed (Participants) | 40 | 44
  Pain or discomfort during sex - period 3 | 0.38 (1.04) | 0.12 (0.60)
  Ringing in ears or noise intolerance - period 1 | 0.73 (1.34) | 0.61 (1.26)
  Ringing in ears or noise intolerance - period 2: number analyzed (Participants) | 42 | 46
  Ringing in ears or noise intolerance - period 2 | 0.58 (1.12) | 0.67 (1.31)
  Ringing in ears or noise intolerance - period 3: number analyzed (Participants) | 40 | 44
  Ringing in ears or noise intolerance - period 3 | 0.61 (1.30) | 0.60 (1.19)
  Shortness of breath - period 1 | 0.86 (1.37) | 0.94 (1.41)
  Shortness of breath - period 2: number analyzed (Participants) | 42 | 46
  Shortness of breath - period 2 | 1.00 (1.48) | 0.81 (1.39)
  Shortness of breath - period 3: number analyzed (Participants) | 40 | 44
  Shortness of breath - period 3 | 0.73 (1.29) | 0.72 (1.30)
  Speech difficulties - period 1 | 0.27 (0.87) | 0.34 (0.97)
  Speech difficulties - period 2: number analyzed (Participants) | 42 | 46
  Speech difficulties - period 2 | 0.34 (0.95) | 0.25 (0.82)
  Speech difficulties - period 3: number analyzed (Participants) | 40 | 44
  Speech difficulties - period 3 | 0.42 (1.06) | 0.21 (0.73)
  Difficulty staying asleep - period 1 | 1.44 (1.61) | 1.48 (1.66)
  Difficulty staying asleep - period 2: number analyzed (Participants) | 42 | 46
  Difficulty staying asleep - period 2 | 1.49 (1.73) | 1.19 (1.61)
  Difficulty staying asleep - period 3: number analyzed (Participants) | 40 | 44
  Difficulty staying asleep - period 3 | 1.53 (1.69) | 1.22 (1.64)
  Difficulty with urination - period 1 | 0.45 (1.09) | 0.32 (0.96)
  Difficulty with urination - period 2: number analyzed (Participants) | 42 | 46
  Difficulty with urination - period 2 | 0.55 (1.19) | 0.28 (0.89)
  Difficulty with urination - period 3: number analyzed (Participants) | 40 | 44
  Difficulty with urination - period 3 | 0.48 (1.05) | 0.30 (0.91)
  Nausea or vomiting - period 1 | 0.56 (1.16) | 0.27 (0.80)
  Nausea or vomiting - period 2: number analyzed (Participants) | 42 | 46
  Nausea or vomiting - period 2 | 0.46 (1.08) | 0.34 (0.95)
  Nausea or vomiting - period 3: number analyzed (Participants) | 40 | 44
  Nausea or vomiting - period 3 | 0.41 (1.02) | 0.19 (0.69)
  Unplanned changes in weight - period 1 | 0.71 (1.39) | 0.90 (1.52)
  Unplanned changes in weight - period 2: number analyzed (Participants) | 42 | 46
  Unplanned changes in weight - period 2 | 0.41 (1.02) | 0.19 (0.69)
  Unplanned changes in weight - period 3: number analyzed (Participants) | 40 | 44
  Unplanned changes in weight - period 3 | 0.73 (1.38) | 0.57 (1.22)
Statistical Analysis 1: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "neuropathy" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "neuropathy" score from period 1 to period 2 between the two arms; p = 0.02, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.32 — The parameter was estimated using a difference in change in "neuropathy" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 2: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "problems maintaining an erection" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "problems maintaining an erection" score from period 1 to period 2 between the two arms; p = 0.11, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.29 — The parameter was estimated using a difference in change in "problems maintaining an erection" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 3: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "dry mouth" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "dry mouth" score from period 1 to period 2 between the two arms; p = 0.02, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.29 — The parameter was estimated using a difference in change in "dry mouth" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 4: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "ringing in ear" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "ringing in ear" score from period 1 to period 2 between the two arms; p = 0.01, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.29 — The parameter was estimated using a difference in change in "ringing in ear" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 5: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "vomit" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "vomit" score from period 1 to period 2 between the two arms; p = 0.01, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.28 — The parameter was estimated using a difference in change in "vomit" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 6: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "dry eyes" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "dry eyes" score from period 1 to period 2 between the two arms; p = 0.02, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.24 — The parameter was estimated using a difference in change in "dry eyes" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 7: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "heartburn" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "heartburn" score from period 1 to period 2 between the two arms; p = 0.11, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.19 — The parameter was estimated using a difference in change in "heartburn" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 8: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "diarrhea" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "diarrhea" score from period 1 to period 2 between the two arms; p = 0.21, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.16 — The parameter was estimated using a difference in change in "diarrhea" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 9: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "constipation" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "constipation" score from period 1 to period 2 between the two arms; p = 0.33, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.14 — The parameter was estimated using a difference in change in "constipation" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 10: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "appetite change" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "appetite change" score from period 1 to period 2 between the two arms; p = 0.46, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.10 — The parameter was estimated using a difference in change in "appetite change" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 11: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "difficulty remembering" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "difficulty remembering" score from period 1 to period 2 between the two arms; p = 0.46, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.10 — The parameter was estimated using a difference in change in "difficulty remembering" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 12: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "fatigue" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "fatigue" score from period 1 to period 2 between the two arms; p = 0.58, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.07 — The parameter was estimated using a difference in change in "fatigue" score from period 1 to period 2 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 13: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "cough" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "cough" score from period 1 to period 2 between the two arms; p = 0.92, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.01 — The parameter was estimated using a difference in change in "cough" score from period 1 to period 2 between the two arms
Statistical Analysis 14: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "urination" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "urination" score from period 1 to period 2 between the two arms; p = 0.84, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.02 — The parameter was estimated using a difference in change in "urination" score from period 1 to period 2 between the two arms
Statistical Analysis 15: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "clumsy" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "clumsy" score from period 1 to period 2 between the two arms; p = 0.83, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.03 — The parameter was estimated using a difference in change in "clumsy" score from period 1 to period 2 between the two arms
Statistical Analysis 16: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "fever" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "fever" score from period 1 to period 2 between the two arms; p = 0.72, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.04 — The parameter was estimated using a difference in change in "fever" score from period 1 to period 2 between the two arms
Statistical Analysis 17: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "pain during sex" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "pain during sex" score from period 1 to period 2 between the two arms; p = 0.48, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.06 — The parameter was estimated using a difference in change in "pain during sex" score from period 1 to period 2 between the two arms
Statistical Analysis 18: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "dizziness" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "dizziness" score from period 1 to period 2 between the two arms; p = 0.54, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.08 — The parameter was estimated using a difference in change in "dizziness" score from period 1 to period 2 between the two arms
Statistical Analysis 19: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "muscle aches" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "muscle aches" score from period 1 to period 2 between the two arms; p = 0.56, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.09 — The parameter was estimated using a difference in change in "muscle aches" score from period 1 to period 2 between the two arms
Statistical Analysis 20: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "speech difficulties" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "speech difficulties" score from period 1 to period 2 between the two arms; p = 0.22, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.10 — The parameter was estimated using a difference in change in "speech difficulties" score from period 1 to period 2 between the two arms
Statistical Analysis 21: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "decreased sex drive" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "decreased sex drive" score from period 1 to period 2 between the two arms; p = 0.40, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.11 — The parameter was estimated using a difference in change in "decreased sex drive" score from period 1 to period 2 between the two arms
Statistical Analysis 22: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "anxiety" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "anxiety" score from period 1 to period 2 between the two arms; p = 0.35, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.13 — The parameter was estimated using a difference in change in "anxiety" score from period 1 to period 2 between the two arms
Statistical Analysis 23: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "difficulty concentrating" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "difficulty concentrating" score from period 1 to period 2 between the two arms; p = 0.11, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.17 — The parameter was estimated using a difference in change in "difficulty concentrating" score from period 1 to period 2 between the two arms
Statistical Analysis 24: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "shortness of breath" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "shortness of breath" score from period 1 to period 2 between the two arms; p = 0.11, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.20 — The parameter was estimated using a difference in change in "shortness of breath" score from period 1 to period 2 between the two arms
Statistical Analysis 25: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "difficulty falling asleep" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "difficulty falling asleep" score from period 1 to period 2 between the two arms; p = 0.15, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.20 — The parameter was estimated using a difference in change in "difficulty falling asleep" score from period 1 to period 2 between the two arms
Statistical Analysis 26: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "unplanned changes in weight" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "unplanned changes in weight" score from period 1 to period 2 between the two arms; p = 0.08, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.22 — The parameter was estimated using a difference in change in "unplanned changes in weight" score from period 1 to period 2 between the two arms
Statistical Analysis 27: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "depression" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "depression" score from period 1 to period 2 between the two arms; p = 0.02, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.34 — The parameter was estimated using a difference in change in "depression" score from period 1 to period 2 between the two arms
Statistical Analysis 28: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "difficulty staying asleep" score from period 1 to period 2 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "difficulty staying asleep" score from period 1 to period 2 between the two arms; p = 0.01, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.36 — The parameter was estimated using a difference in change in "difficulty staying asleep" score from period 1 to period 2 between the two arms
Statistical Analysis 29: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "dry mouth" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "dry mouth" score from period 1 to period 3 between the two arms; p = 0.08, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.27 — The parameter was estimated using a difference in change in "dry mouth" score from period 1 to period 3 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 30: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "ringing in ear" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "ringing in ear" score from period 1 to period 3 between the two arms; p = 0.08, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.24 — The parameter was estimated using a difference in change in "ringing in ear" score from period 1 to period 3 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 31: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "dry eyes" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "dry eyes" score from period 1 to period 3 between the two arms; p = 0.08, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.24 — The parameter was estimated using a difference in change in "dry eyes" score from period 1 to period 3 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 32: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "maintaining an erection" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "maintaining an erection" score from period 1 to period 3 between the two arms; p = 0.71, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.13 — The parameter was estimated using a difference in change in "maintaining an erection" score from period 1 to period 3 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 33: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "vomit" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "vomit" score from period 1 to period 3 between the two arms; p = 0.41, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.11 — The parameter was estimated using a difference in change in "vomit" score from period 1 to period 3 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 34: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "neuropathy" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "neuropathy" score from period 1 to period 3 between the two arms; p = 0.84, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.08 — The parameter was estimated using a difference in change in "neuropathy" score from period 1 to period 3 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 35: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "urination" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "urination" score from period 1 to period 3 between the two arms; p = 0.71, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.07 — The parameter was estimated using a difference in change in "urination" score from period 1 to period 3 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 36: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "appetite change" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "appetite change" score from period 1 to period 3 between the two arms; p = 0.88, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.05 — The parameter was estimated using a difference in change in "appetite change" score from period 1 to period 3 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 37: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "shortness of breath" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "shortness of breath" score from period 1 to period 3 between the two arms; p = 0.93, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.03 — The parameter was estimated using a difference in change in "shortness of breath" score from period 1 to period 3 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 38: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "difficulty remembering" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "difficulty remembering" score from period 1 to period 3 between the two arms; p = 0.93, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.03 — The parameter was estimated using a difference in change in "difficulty remembering" score from period 1 to period 3 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 39: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "muscle aches" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "muscle aches" score from period 1 to period 3 between the two arms; p = 0.94, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.03 — The parameter was estimated using a difference in change in "muscle aches" score from period 1 to period 3 between the two arms. Negative estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 40: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "diarrhea" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "diarrhea" score from period 1 to period 3 between the two arms; p = 0.97, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.004 — The parameter was estimated using a difference in change in "diarrhea" score from period 1 to period 3 between the two arms
Statistical Analysis 41: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "fatigue" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "fatigue" score from period 1 to period 3 between the two arms; p = 0.95, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.01 — The parameter was estimated using a difference in change in "fatigue" score from period 1 to period 3 between the two arms
Statistical Analysis 42: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "anxiety" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "anxiety" score from period 1 to period 3 between the two arms; p = 0.95, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.01 — The parameter was estimated using a difference in change in "anxiety" score from period 1 to period 3 between the two arms
Statistical Analysis 43: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "constipation" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "constipation" score from period 1 to period 3 between the two arms; p = 0.93, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.03 — The parameter was estimated using a difference in change in "constipation" score from period 1 to period 3 between the two arms
Statistical Analysis 44: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "fever" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "fever" score from period 1 to period 3 between the two arms; p = 0.84, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.06 — The parameter was estimated using a difference in change in "fever" score from period 1 to period 3 between the two arms
Statistical Analysis 45: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "cough" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "cough" score from period 1 to period 3 between the two arms; p = 0.84, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.07 — The parameter was estimated using a difference in change in "cough" score from period 1 to period 3 between the two arms
Statistical Analysis 46: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "heartburn" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "heartburn" score from period 1 to period 3 between the two arms; p = 0.54, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.11 — The parameter was estimated using a difference in change in "heartburn" score from period 1 to period 3 between the two arms
Statistical Analysis 47: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "pain during sex" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "pain during sex" score from period 1 to period 3 between the two arms; p = 0.13, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.14 — The parameter was estimated using a difference in change in "pain during sex" score from period 1 to period 3 between the two arms
Statistical Analysis 48: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "clumsy" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "clumsy" score from period 1 to period 3 between the two arms; p = 0.18, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.18 — The parameter was estimated using a difference in change in "clumsy" score from period 1 to period 3 between the two arms
Statistical Analysis 49: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "difficulty falling asleep" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "difficulty falling asleep" score from period 1 to period 3 between the two arms; p = 0.29, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.19 — The parameter was estimated using a difference in change in "difficulty falling asleep" score from period 1 to period 3 between the two arms
Statistical Analysis 50: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "difficulty concentrating" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "difficulty concentrating" score from period 1 to period 3 between the two arms; p = 0.12, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.20 — The parameter was estimated using a difference in change in "difficulty concentrating" score from period 1 to period 3 between the two arms
Statistical Analysis 51: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "decreased sex drive" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "decreased sex drive" score from period 1 to period 3 between the two arms; p = 0.10, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.24 — The parameter was estimated using a difference in change in "decreased sex drive" score from period 1 to period 3 between the two arms
Statistical Analysis 52: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "speech difficulties" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "speech difficulties" score from period 1 to period 3 between the two arms; p = 0.01, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.25 — The parameter was estimated using a difference in change in "speech difficulties" score from period 1 to period 3 between the two arms
Statistical Analysis 53: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "unplanned changes in weight" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "unplanned changes in weight" score from period 1 to period 3 between the two arms; p = 0.08, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.26 — The parameter was estimated using a difference in change in "unplanned changes in weight" score from period 1 to period 3 between the two arms
Statistical Analysis 54: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "dizziness" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "dizziness" score from period 1 to period 3 between the two arms; p = 0.08, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.27 — The parameter was estimated using a difference in change in "dizziness" score from period 1 to period 3 between the two arms
Statistical Analysis 55: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "difficulty staying asleep" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "difficulty staying asleep" score from period 1 to period 3 between the two arms; p = 0.09, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.27 — The parameter was estimated using a difference in change in "difficulty staying asleep" score from period 1 to period 3 between the two arms
Statistical Analysis 56: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in mean "depression" score from period 1 to period 3 between the two arms; Test type: Superiority — Linear mixed models to test difference in mean "depression" score from period 1 to period 3 between the two arms; p = 0.05, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.38 — The parameter was estimated using a difference in change in "depression" score from period 1 to period 3 between the two arms

2. Secondary Outcome: Score on Patient-Reported Outcomes Measurement Information System® (PROMIS)-29
Description: The PROMIS-29 includes seven health related quality of life domains (Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, and Pain), and the pain domain has two subdomains (interference and intensity). Each of the 7 domains has four 5-level items (i.e., 16 decrements each). In addition to these items, pain intensity is assessed using a single 11-point numeric rating scale anchored between no pain (0) and worse imaginable pain. Raw scores, except pain intensity, are transformed using the T-score metric based on the item response theory calibrations in which scores have a mean of 50 and standard deviation of 10 for the general population in the US. T-scores can be estimated using scoring tables listed in the PROMIS manuals. A higher PROMIS T-score implies more of the concept being measured; i.e., a higher PROMIS score on physical function indicates better functioning, whereas a higher score on depression indicates more severe depressive symptoms.
Time Frame: Baseline, 3 months, and 6 months
Population: Not all participants completed the scale at 3 months and 6 months because they did not show up to their 3-month and 6-month follow-up visit. Some participants also did not answer all of the questions within the scale to produce a valid t-score, and were thus excluded from the analysis.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 50 | 50
T-Score
  Physical Function at Baseline: number analyzed (Participants) | 50 | 49
  Physical Function at Baseline | 43.79 (9.28) | 41.43 (8.18)
  Physical Function at 3 months: number analyzed (Participants) | 43 | 46
  Physical Function at 3 months | 45.37 (9.09) | 41.98 (8.46)
  Physical Function at 6 months: number analyzed (Participants) | 41 | 45
  Physical Function at 6 months | 44.35 (9.29) | 41.63 (7.43)
  Anxiety at Baseline | 56.28 (9.45) | 55.56 (9.67)
  Anxiety at 3 months: number analyzed (Participants) | 43 | 46
  Anxiety at 3 months | 54.88 (8.29) | 55.03 (9.02)
  Anxiety at 6 months: number analyzed (Participants) | 41 | 45
  Anxiety at 6 months | 44.35 (9.29) | 53.32 (9.46)
  Depression at Baseline | 53.58 (8.56) | 53.32 (10.11)
  Depression at 3 months: number analyzed (Participants) | 43 | 46
  Depression at 3 months | 52.12 (8.64) | 52.52 (10.02)
  Depression at 6 months: number analyzed (Participants) | 41 | 44
  Depression at 6 months | 52.62 (7.89) | 52.34 (8.54)
  Fatigue at Baseline | 53.81 (9.40) | 52.99 (9.00)
  Fatigue at 3 months: number analyzed (Participants) | 43 | 46
  Fatigue at 3 months | 51.75 (9.93) | 52.63 (10.21)
  Fatigue at 6 months: number analyzed (Participants) | 41 | 45
  Fatigue at 6 months | 54.23 (9.28) | 51.46 (8.45)
  Sleep Disturbance at Baseline | 54.98 (8.79) | 54.66 (8.63)
  Sleep Disturbance at 3 months: number analyzed (Participants) | 43 | 46
  Sleep Disturbance at 3 months | 52.69 (8.95) | 51.52 (9.58)
  Sleep Disturbance at 6 months: number analyzed (Participants) | 41 | 45
  Sleep Disturbance at 6 months | 52.54 (8.28) | 50.29 (9.30)
  Satisfaction with Social Role at Baseline | 47.31 (9.97) | 45.05 (8.64)
  Satisfaction with Social Role at 3 months: number analyzed (Participants) | 43 | 46
  Satisfaction with Social Role at 3 months | 48.00 (9.88) | 45.99 (9.52)
  Satisfaction with Social Role at 6 months: number analyzed (Participants) | 41 | 45
  Satisfaction with Social Role at 6 months | 48.47 (8.47) | 46.15 (8.10)
  Pain Interference at Baseline | 59.12 (7.70) | 59.56 (8.59)
  Pain Interference at 3 months: number analyzed (Participants) | 43 | 46
  Pain Interference at 3 months | 56.56 (10.73) | 57.52 (9.45)
  Pain Interference at 6 months: number analyzed (Participants) | 41 | 45
  Pain Interference at 6 months | 57.43 (9.53) | 56.94 (7.28)
Statistical Analysis 1: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Fatigue PROMIS T-score from baseline to 3 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Fatigue PROMIS T-score from baseline to 3 months between two arms; p = 0.83, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -2.09 — The parameter was estimated using a difference in change in Fatigue PROMIS T-score from baseline to 3 months between two arms
Statistical Analysis 2: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Anxiety PROMIS T-score from baseline to 3 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Anxiety PROMIS T-score from baseline to 3 months between two arms; p = 0.83, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.94 — The parameter was estimated using a difference in change in Anxiety PROMIS T-score from baseline to 3 months between two arms
Statistical Analysis 3: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Depression PROMIS T-score from baseline to 3 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Depression PROMIS T-score from baseline to 3 months between two arms; p = 0.83, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.79 — The parameter was estimated using a difference in change in Depression PROMIS T-score from baseline to 3 months between two arms
Statistical Analysis 4: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Pain Interference PROMIS T-score from baseline to 3 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Pain Interference PROMIS T-score from baseline to 3 months between two arms; p = 0.83, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.78 — The parameter was estimated using a difference in change in Pain Interference PROMIS T-score from baseline to 3 months between two arms
Statistical Analysis 5: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Satisfaction with Social Role PROMIS T-score from baseline to 3 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Satisfaction with Social Role PROMIS T-score from baseline to 3 months between two arms; p = 0.98, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.04 — The parameter was estimated using a difference in change in Satisfaction with Social Role PROMIS T-score from baseline to 3 months between two arms. Positive estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 6: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Physical Function PROMIS T-score from baseline to 3 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Physical Function PROMIS T-score from baseline to 3 months between two arms; p = 0.83, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.55 — The parameter was estimated using a difference in change in Physical Function PROMIS T-score from baseline to 3 months between two arms. Positive estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 7: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Sleep Disturbance PROMIS T-score from baseline to 3 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Sleep Disturbance PROMIS T-score from baseline to 3 months between two arms; p = 0.83, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.84 — The parameter was estimated using a difference in change in Sleep Disturbance PROMIS T-score from baseline to 3 months between two arms. Positive estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 8: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Physical Function PROMIS T-score from baseline to 6 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Physical Function PROMIS T-score from baseline to 6 months between two arms; p = 0.96, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = -0.43 — The parameter was estimated using a difference in change in Physical Function PROMIS T-score from baseline to 6 months between two arms
Statistical Analysis 9: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Depression PROMIS T-score from baseline to 6 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Depression PROMIS T-score from baseline to 6 months between two arms; p = 0.96, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.07 — The parameter was estimated using a difference in change in Depression PROMIS T-score from baseline to 6 months between two arms. Positive estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 10: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Satisfaction with Social Role PROMIS T-score from baseline to 6 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Satisfaction with Social Role PROMIS T-score from baseline to 6 months between two arms; p = 0.96, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.23; The parameter was estimated using a difference in change in Satisfaction with Social Role PROMIS T-score from baseline to 6 months between two arms. Positive estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 11: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Anxiety PROMIS T-score from baseline to 6 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Anxiety PROMIS T-score from baseline to 6 months between two arms; p = 0.96, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 0.77 — The parameter was estimated using a difference in change in Anxiety PROMIS T-score from baseline to 6 months between two arms. Positive estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 12: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Pain Interference PROMIS T-score from baseline to 6 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Pain Interference PROMIS T-score from baseline to 6 months between two arms; p = 0.96, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 1.05 — The parameter was estimated using a difference in change in Pain Interference PROMIS T-score from baseline to 6 months between two arms. Positive estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 13: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Fatigue PROMIS T-score from baseline to 6 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Fatigue PROMIS T-score from baseline to 6 months between two arms; p = 0.96, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 1.50 — The parameter was estimated using a difference in change in Fatigue PROMIS T-score from baseline to 6 months between two arms. Positive estimation parameter value indicates intervention arm better than control arm
Statistical Analysis 14: Comparison: Intervention vs Control; The null hypothesis is that there is no difference in change in Sleep Disturbance PROMIS T-score from baseline to 6 months between two arms; Test type: Superiority — Linear mixed models to test difference in mean score of Sleep Disturbance PROMIS T-score from baseline to 6 months between two arms; p = 0.64, Linear mixed model — Calculated p-value given the null-hypothesis. P value was adjusted for multiple-test with a false discovery rate (FDR); Difference in Change = 2.04 — The parameter was estimated using a difference in change in Sleep Disturbance PROMIS T-score from baseline to 6 months between two arms. Positive estimation parameter value indicates intervention arm better than control arm

3. Other Pre Specified Outcome: Change in Score on SF-12
Description: 12-Item Medical Outcomes Study Short Form (SF-12) is a health survey to measure health-related quality of life.
Time Frame: 3 months and 6 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Score on Engagement With Health Care Provider Scale
Description: Engagement with Health Care Provide scale is a 13-item scale in which subjects rate their interactions with their health care providers on a four-point scale with 1=always true and 4=never true. A total score can be calculated to create a possible range of 13-52. A low score (closer to 13) indicates greater provider engagement between the patient and provider.
Time Frame: Baseline, 3 months, and 6 months
Population: Not all participants completed the scale at 3 months and 6 months because they did not show up to their 3-month and 6-month follow-up visit. Some participants also did not answer all of the questions within the scale to produce a score between 13 and 52, and were thus excluded from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 50 | 50
score on a scale
  Score at Baseline: number analyzed (Participants) | 50 | 47
  Score at Baseline | 17.78 (8.07) | 17.13 (6.52)
  Score at 3-months: number analyzed (Participants) | 42 | 43
  Score at 3-months | 20.17 (8.68) | 17.33 (5.43)
  Score at 6-months: number analyzed (Participants) | 39 | 44
  Score at 6-months | 18.05 (7.72) | 18.70 (8.02)

5. Other Pre Specified Outcome: Score of the VAS
Description: The Visual Analogue Scale (VAS) measures adherence to antiretroviral therapy (ART). VAS asks subjects to indicate a point on a line that shows their best guess about how much of each drug they have taken. 0% means they have taken no drug, 50% means they have taken half their drugs, and 100% means they have taken every single dose.
Time Frame: Baseline, 3 months, and 6 months
Population: Not all participants completed the scale at 3 months and 6 months because they did not show up to their 3-month and 6-month follow-up visit. Some participants also did not answer the question and left it blank, thus excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage of medication
Arm/Group | Intervention | Control
Number analyzed (Participants) | 50 | 50
percentage of medication
  Baseline VAS Score: number analyzed (Participants) | 45 | 48
  Baseline VAS Score | 88.49 (17.34) | 83.91 (26.45)
  3-month VAS Score: number analyzed (Participants) | 38 | 44
  3-month VAS Score | 86.89 (24.43) | 87.30 (20.99)
  6-month VAS score: number analyzed (Participants) | 40 | 42
  6-month VAS score | 86.88 (21.49) | 88.63 (20.45)

6. Other Pre Specified Outcome: Score on Fried's Frailty Phenotype
Description: Fried's frailty phenotype is a combination of five scores: weight loss in the last year, exhaustion, physical activity, walk time for a 15 foot interval, and grip strength. The frailty condition is defined as meeting the definition of frailty for at least 3 of the listed scores.
Time Frame: Baseline, 3 months, and 6 months
Population: Not all participants showed up to their 3-month and 6-month follow-up visit and therefore did not complete any of the frailty measures. These individuals were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 50 | 50
Participants
  Frail at Baseline | 25 | 26
  Frail at 3 months: number analyzed (Participants) | 43 | 46
  Frail at 3 months | 19 | 21
  Frail at 6 months: number analyzed (Participants) | 41 | 45
  Frail at 6 months | 17 | 17

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 1 year time period.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT03182738/Prot_SAP_000.pdf